CLINICAL TRIAL: NCT05355441
Title: Pain Multidisciplinar Intervention Effect in Major Trauma Patients. Does it Improve the Quality of Life?
Brief Title: Pain Multidisciplinar Intervention in Major Trauma Patients
Status: Completed | Type: Observational
Sponsor: Nuria Llorach-Perucho (Other)
Collaborators: Corporacion Parc Tauli (Other)
Responsible Party: Sponsor-Investigator, Nuria Llorach-Perucho, Principal Investigator, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Other Study IDs: DOLOTRAU
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Trauma; Chronic Pain; Psychological Trauma
MeSH Terms: conditions — Wounds and Injuries; Chronic Pain; Psychological Trauma | interventions — Acetaminophen; Ibuprofen; Tramadol; Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multidisciplinar pain treatment patients: Major trauma patients with moderate, severe or incapacitating pain will be referred to consultation specialized in chronic pain and psychology. Patients will be evaluated, in terms of quality of life, before and after the treatment.
  Interventions: Drug: Paracetamol; Drug: Ibuprofen 600 mg; Drug: Tramadol; Drug: Morphine

INTERVENTIONS:
Drug: Paracetamol — Routine clinical practice treatments recommended by the medical team involved
  Other Names: Psychological drugs
Drug: Ibuprofen 600 mg — Routine clinical practice treatments recommended by the medical team involved
  Other Names: Psychological drugs
Drug: Tramadol — Routine clinical practice treatments recommended by the medical team involved
  Other Names: Psychological drugs
Drug: Morphine — Routine clinical practice treatments recommended by the medical team involved
  Other Names: Psychological drugs

SUMMARY:
In Spain, major trauma continues to be the leading cause of death among young people. However, mortality rates represent only a relatively small part of the impact of trauma injuries on the health of the population. Pain and anxiety are two of the most poorly controlled factors that have a huge impact on a patient's quality of life.The type of therapy that has been shown to be most effective in treating post-traumatic pain is one that involves different specialists, given its multicausality, care should be multidisciplinary.

This investigation project consists in an observational study performed by a multidisciplinary team in our center. Major trauma patients with moderate, severe or incapacitating pain will be referred to consultations specialized in chronic pain and psychology. One year after the trauma, patients will be evaluated in terms of quality of life.

The aim of this study is to determinate the impact that multidisciplinary treatment of post-traumatic pain has on the perception of quality of life in severely injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Major trauma patients with moderate, severe or incapacitating pain (according to EQ-5D-5L scale).

Exclusion Criteria:

* Death in the first 30 days after the trauma.
* Transferred to another center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major trauma patients with moderate, severe or incapacitating pain after hospital discharge.
  Major trauma patients are defined as trauma patients that require an admission on the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Perception of quality of life according to EQ-5D-5L questionnaire | 1 year
  Perception of quality of life after multidisciplinar pain intervention according to European Quality of Life 5 Dimensions (EQ-5D-5L) questionnaire (0-100; poor health - good health)

SECONDARY OUTCOMES:
Type of pain according to EVA scale | 1 year
  Type and severity of pain according to EVA (visual pain scale: 0-10; no pain to lot of pain)
Type of treatments requiered | 1 year
  Type of treatments required (anti inflammatory, opioid, adjuvants, invasive procedures)
Number of visits requiered in chronic pain and psychologic specialists | 1 year
  Number of visits requiered in chronic pain and psychologic specialist

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Llorach-Perucho, MD, Principal Investigator — Corporacion Parc Tauli; Salvador Navarro-Soto, MD, PhD, Study Director — Corporacion Parc Tauli; Heura Llaquet-Bayo, MD, PhD, Study Director — Corporacion Parc Tauli
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain